CLINICAL TRIAL: NCT01649583
Title: A Feasibility Study to Evaluate Use of the Jaw Dynasplint System to Prevent Trismus in Patients With Head and Neck Cancer Receiving Primary or Adjuvant Radiation-Based Therapy
Brief Title: Feasibility Study of Dynasplint to Prevent Trismus in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Zatarain, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 120727
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Trismus; Head and Neck Cancer
MeSH Terms: conditions — Trismus; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaw Dynasplint System (Experimental)
  Interventions: Device: Jaw Dynasplint System
- Control Arm (No Intervention)

INTERVENTIONS:
Device: Jaw Dynasplint System — Patients on the intervention arm will wear the Jaw Dynasplint® System for 30 minutes, 3 times per day each day during the cancer treatment period and for the first 3 months after primary or adjuvant based-radiation treatment (recovery period) is completed. Patients will maintain a daily patient log indicating the amount of time they used the Jaw Dynasplint® System.
  Other Names: Trismus Dynasplint; Mechanical Stretching Device
  Arms: Jaw Dynasplint System

SUMMARY:
The purpose of this study is to see if use of a device called the Jaw Dynasplint® System can be used during and immediately after cancer treatment. The Dynasplint® is a stretching device that is used to treat joint stiffness and limited range of motion in the jaw. The device is currently approved for treatment of trismus once it has developed. This study will investigate the use of the device during and immediately after cancer treatment to prevent trismus.

DETAILED DESCRIPTION:
Data suggest that early intervention with mechanical stretching devices for head and neck cancer patients undergoing curative therapy maximizes their effectiveness in the treatment of trismus. That being said, treatment for trismus typically begins after head and neck cancer patients are found to have moderate to severe reduction in jaw range of motion. Typically, clinicians will begin therapy when the IID is 3.0 cm or less. A subset of head and neck cancer patients will develop severe or rapidly progressive trismus that will fail to respond to treatment. In this cohort, trismus may lead to permanent, severe morbidity. It may be hypothesized that preventative strategies that encourage routine stretching during and immediately after the completion of cancer therapy may prevent or minimize trismus. No studies have examined the prophylactic use of the Jaw Dynasplint® System during cancer treatment.

Furthermore, it is not known whether patients can tolerate wearing a mechanical stretching device during treatment. The investigators would like to test the hypothesis that: 1) preventive use of a mechanical stretching device during cancer treatment and early recovery is feasible, and 2) preventive use of a mechanical stretching device will result in a marked decrease in the incidence and severity of trismus in patients undergoing primary or adjuvant radiation therapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven head and neck cancer
2. Planned primary or adjuvant radiation treatment with 50cGy or greater delivered to a total volume of at least 2cc to the muscles of mastication, unilaterally or bilaterally, over the entire course of radiation treatment
3. Patients receiving induction or concurrent chemotherapy
4. Baseline interincisoral distance > 35 mm
5. Willing and able to provide informed consent
6. Sufficient manual dexterity to utilize the device
7. All participants must be at least 21 years of age

Exclusion Criteria:

1. Patients with collagen vascular disorders that may predispose to radiation fibrosis
2. Patients with oral health issues that would preclude use of the device as identified during a pre-radiation dental evaluation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of use of a Dynasplint during chemoradiation for head and neck cancer patients | 2 years
  Feasibility will be measured based on patient compliance, adverse events, and barriers to use of the Jaw Dynasplint® System.

SECONDARY OUTCOMES:
Preliminary Efficacy Data on Prevention of Trismus | 2 years
  Interincisoral distance (IID) will be the primary measure of efficacy. Any patient who develops IID of 30 mm or less will be considered to have clinically significant trismus. The incidence of trismus will be compared between the intervention arm (Arm 1) and the standard of care arm (Arm 2).

OTHER OUTCOMES:
Symptom Burden of Patients with Trismus | 2 years
  Patient reported outcome data will be collected via questionnaires including, the Vanderbilt Head and Neck Symptom Survey plus General Symptom Survey version 2.0 (VHNSS v2.0 plus GSS), and the Mandibular Function Impairment Questionnaire (MFIQ). This patient reported outcome data will be collected in order to identify correlations between trismus and symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren A Zatarain, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States